CLINICAL TRIAL: NCT06073730
Title: Department of Hematology, The Second Affiliated Hospital of Kunming Medical University.
Brief Title: Comparison of the Efficacy and Safety of Venetoclax in Combination With 3 Days Decitabine (DEC3-VEN) vs. Venetoclax in Combination With Azacitidine (VIALE-A) in the Treatment of Elderly Patients or Unfit, New-diagnosis Acute Myeloid Leukemia Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, ZePing Zhou, Dr., The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEN-PJ-KE-2023-223
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Elderly AML Patients; Unfit, New-diagnosis AML; Acute Myeloid Leukemia; Venetoclax; Decitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Sorafenib; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venetoclax in combination with Decitabine (+-sorafenib) (Experimental): Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-14 Decitabine (DEC) 20mg/m2/q8h, d4-6 (infusion time >2h) Sorafenib 600mg/d, d8-14 (FLT3/ITD mutation positive patients)
  Interventions: Procedure: Experimental: Venetoclax in combination with Decitabine (+-sorafenib)
- Standard dose of Venetoclax + Azacitidine (Active Comparator): Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-28 Azacitidine (AZA) 75mg/m2/d, d3-9
  Interventions: Procedure: Active Comparator: Standard dose of Venetoclax + Azacitidine

INTERVENTIONS:
Procedure: Experimental: Venetoclax in combination with Decitabine (+-sorafenib) — Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-14 Decitabine (DEC) 20mg/m2/q8h, d4-6 (infusion time >2h) Sorafenib 600mg/d, d8-14 (FLT3/ITD mutation positive patients)
  Other Names: DEC3-VEN
  Arms: Venetoclax in combination with Decitabine (+-sorafenib)
Procedure: Active Comparator: Standard dose of Venetoclax + Azacitidine — Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-28 Azacitidine (AZA) 75mg/m2/d, d3-9
  Arms: Standard dose of Venetoclax + Azacitidine

SUMMARY:
Combining the results of previous studies and based on the clinical practice in our center, we designed the Venetoclax in combination with 3days-Decitabine regimen for induction therapy in elderly or unfit AML patients with a primary diagnosis, and set Venetoclax in combination with Azacitidine (VIALE-A) as a control group to compare the efficacy and safety and to provide evidence for the optimal selection of the clinical treatment regimen.

PRIMARY ENDPOINT: To assess whether Venetoclax in combination with 3 days-diascitabine versus standard dose Venetoclax in combination with azacitidine improves event-free survival (EFS) in elderly or adult patients with unfit AML during the maximum follow-up period. Event-free survival was defined as the absence of events such as treatment failure, intolerance withdrawal, all-cause death, or achievement of CR or CRi, or relapse after MLFS, whichever occurred first, between patients' randomization and the maximum follow-up period. Treatment failure was defined as failure to achieve CR or CRi, MLFS after 2 courses of induction therapy.

DETAILED DESCRIPTION:
Induction therapy regimen:

A: Experimental group: Venetoclax in combination with Decitabine (+-sorafenib) Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-14 Decitabine (DEC) 20mg/m2/q8h, d4-6 (infusion time >2h) Sorafenib 600mg/d, d8-14 (FLT3/ITD mutation positive patients) B: Control: standard dose of Venetoclax + Azacitidine Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-28 Azacitidine (AZA) 75mg/m2/d, d3-9

Post-remission treatment regimen:

A: Experimental group: Venetoclax combined with Decitabine Venetoclax (VEN ) 400mg/d, d1-7 Decitabine (DEC) 20mg/m2/q8h, d2-3 (this regimen is repeated every 4-6 weeks) B: Control Group: Venetoclax combined with Azacitidine Venetoclax (VEN ) 100mg d1, 200mg d2, 400mg/d d3-28 Azacitidine (AZA) 75mg/m2/d, d3-9 (this regimen is repeated every 4-6 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Subjects suitable for enrollment in this study must meet all of the following criteria.

  1. meet the World Health Organization diagnostic criteria (WHO2022 criteria) except APL or carry one of the abnormal karyotypes such as t(8;21)/(RUNX1::RUNX1TI), inv(16)(p13.1q22), t(16;16) (p13.1q22), t(16;16)/CBFβ::myh11), etc. Patients with acute myeloid leukemia other than those with one of the abnormal karyotypes such as t(16;16)/CBFβ::myh11
  2. Patients with AML not otherwise classified under the World Health Organization AML classification, except for acute myeloproliferative disorder with myelofibrosis and myeloid sarcoma.
  3. Male or female, A: Elderly patients aged > or = 60 years (unwilling to undergo intense chemotherapy); B: Patients aged > 18 years who are not candidates for standard-dose chemotherapy, defined as those with at least one of the following comorbidities: 1) Eastern Collaborative Oncology Group Physical Conditioning Grading (ECOG) score of 2 or 3; 2) Chronic heart failure (CHF) requiring treatment or with a left ventricular ejection fraction (LVEF) of ≤ 50%; 3) Chronic heart failure (CHF) requiring treatment or with a left ventricular ejection fraction (LVEF) of ≤ 50%. heart failure (CHF) cardiac history or chronic unstable angina; 3) carbon monoxide diffusing capacity (DLCO) ≤65% or forced expiratory volume in 1 second (FEV1) ≤65%; 4) creatinine clearance of ≥30 mL/min to ≤45 mL/min; and 5) any other condition deemed by the investigator to be incompatible with standard-dose chemotherapy must be reviewed with the study chair prior to study enrollment ;
  4. patients have not received prior treatment for AML (except hydroxyurea and Ara-C <1.0 g/d).
  5. Eastern Cooperative Oncology Group Physical Status Assessment (ECOG-PS) score of <=3.
  6. pass the requirements for the following laboratory test indices (performed within 7 days prior to treatment):

  <!-- -->

  1. Aspartate aminotransferase (ALT), alanine aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN), serum bilirubin ≤ 2 x ULN; and serum cardiac enzymes < 2.0 x ULN; unless considered to be leukemic organ involvement.
  2. Creatinine ≥ 30 mL/min, calculated by the Cockcroft Gault formula or measured by 24-hour urine collection.

  7.Subjects of childbearing potential must have a negative pregnancy test result within 72 hours prior to the start of treatment, and participating patients must use contraception during trial treatment and for 3 years after completion of treatment.

  8. life expectancy greater than 2 months. 9. Informed consent must be signed prior to the start of all specific study procedures, either by the patient himself/herself or by a member of his/her immediate family; in view of the patient's condition, if the patient's own signature would not be conducive to the treatment of his/her condition, the informed consent will be signed by the legal guardian or by a member of the patient's immediate family.

Exclusion Criteria:

Subjects may not be enrolled in this study if they meet any of the following criteria:

1. AML with BCR-ABL1; or CML bone marrow acute stage.
2. Treatment-naïve patients (is defined as having received induction chemotherapy in the past, regardless of efficacy).
3. Secondary leukemia (mainly refers to those whose World Health Organization (WHO) AML classification belongs to the subcategory of treatment-related AML and those with a history of prior MDS and/or MPD).
4. concomitant other hematologic diseases (such as hemophilia, myelofibrosis and other investigators considered unsuitable for enrollment; previous blood abnormalities, but ever bone marrow examination except MDS and MPD allowed enrollment).

5、Pregnant or lactating patients. 6, Allergic to any of the drugs involved in this study. 7, Have used strong or moderate CYP7A inducers within 3 days before the start of study treatment.

8, Concomitant malignant tumors of other organs (those requiring treatment). 9, Significantly abnormal hepatic or renal function beyond the enrollment criteria.

10, Active heart disease, defined as one or more of the following:

1. Myocardial infarction less than 6 months from study entry;
2. A history of arrhythmia requiring drug therapy or severe clinical symptoms;
3. Uncontrolled or symptomatic congestive heart failure (> NYHA class 2); 10, patients with severe infectious diseases (untreated tuberculosis, pulmonary aspergillosis), known infection with human immunodeficiency virus (HIV) or active hepatitis B or C.

11. Subjects with evidence of central nervous system leukemia prior to treatment.

Subjects with epilepsy, dementia, or other abnormal mental states that require medication and who are unable to understand or follow the regimen.

13, Conditions that limit oral drug intake or gastrointestinal absorption. 14, Subjects who, in the opinion of the investigator, are not suitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | up to 12 months
  Event-free survival was defined as the absence of events such as treatment failure, intolerance withdrawal, all-cause death, or relapse after achieving CR or CRi, MLFS, whichever occurred first, between patients' randomization and the maximum follow-up period. Treatment failure was defined as failure to achieve CR or CRi, MLFS after 2 courses of induction therapy.

SECONDARY OUTCOMES:
overall survival rate | up to 12 months
  Survival of patients from initiation of treatment to maximum follow-up period
CR/CRi rate | up to 12 months
  CR/CRi rate from initiation of treatment to maximum follow-up period
First course CR/CRi rate | up to 1 months
  CR/CRi rate in patients after receiving the first course of induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University., Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida AM, Prebet T, Itzykson R, Ramos F, Al-Ali H, Shammo J, Pinto R, Maurillo L, Wetzel J, Musto P, Van De Loosdrecht AA, Costa MJ, Esteves S, Burgstaller S, Stauder R, Autzinger EM, Lang A, Krippl P, Geissler D, Falantes JF, Pedro C, Bargay J, Deben G, Garrido A, Bonanad S, Diez-Campelo M, Thepot S, Ades L, Sperr WR, Valent P, Fenaux P, Sekeres MA, Greil R, Pleyer L. Clinical Outcomes of 217 Patients with Acute Erythroleukemia According to Treatment Type and Line: A Retrospective Multinational Study. Int J Mol Sci. 2017 Apr 14;18(4):837. doi: 10.3390/ijms18040837. PMID 28420120
- [Background] Krug U, Buchner T, Berdel WE, Muller-Tidow C. The treatment of elderly patients with acute myeloid leukemia. Dtsch Arztebl Int. 2011 Dec;108(51-52):863-70. doi: 10.3238/arztebl.2011.0863. Epub 2011 Dec 26. PMID 22259641
- [Background] Pettit K, Odenike O. Defining and Treating Older Adults with Acute Myeloid Leukemia Who Are Ineligible for Intensive Therapies. Front Oncol. 2015 Dec 14;5:280. doi: 10.3389/fonc.2015.00280. eCollection 2015. PMID 26697412
- [Background] Kantarjian H, Ravandi F, O'Brien S, Cortes J, Faderl S, Garcia-Manero G, Jabbour E, Wierda W, Kadia T, Pierce S, Shan J, Keating M, Freireich EJ. Intensive chemotherapy does not benefit most older patients (age 70 years or older) with acute myeloid leukemia. Blood. 2010 Nov 25;116(22):4422-9. doi: 10.1182/blood-2010-03-276485. Epub 2010 Jul 28. PMID 20668231
- [Background] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659
- [Background] Kantarjian HM, Thomas XG, Dmoszynska A, Wierzbowska A, Mazur G, Mayer J, Gau JP, Chou WC, Buckstein R, Cermak J, Kuo CY, Oriol A, Ravandi F, Faderl S, Delaunay J, Lysak D, Minden M, Arthur C. Multicenter, randomized, open-label, phase III trial of decitabine versus patient choice, with physician advice, of either supportive care or low-dose cytarabine for the treatment of older patients with newly diagnosed acute myeloid leukemia. J Clin Oncol. 2012 Jul 20;30(21):2670-7. doi: 10.1200/JCO.2011.38.9429. Epub 2012 Jun 11. PMID 22689805
- [Background] Del Poeta G, Venditti A, Del Principe MI, Maurillo L, Buccisano F, Tamburini A, Cox MC, Franchi A, Bruno A, Mazzone C, Panetta P, Suppo G, Masi M, Amadori S. Amount of spontaneous apoptosis detected by Bax/Bcl-2 ratio predicts outcome in acute myeloid leukemia (AML). Blood. 2003 Mar 15;101(6):2125-31. doi: 10.1182/blood-2002-06-1714. Epub 2002 Nov 7. PMID 12424199
- [Background] Mei M, Aldoss I, Marcucci G, Pullarkat V. Hypomethylating agents in combination with venetoclax for acute myeloid leukemia: Update on clinical trial data and practical considerations for use. Am J Hematol. 2019 Mar;94(3):358-362. doi: 10.1002/ajh.25369. Epub 2018 Dec 13. PMID 30499168
- [Background] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] DiNardo CD, Maiti A, Rausch CR, Pemmaraju N, Naqvi K, Daver NG, Kadia TM, Borthakur G, Ohanian M, Alvarado Y, Issa GC, Montalban-Bravo G, Short NJ, Yilmaz M, Bose P, Jabbour EJ, Takahashi K, Burger JA, Garcia-Manero G, Jain N, Kornblau SM, Thompson PA, Estrov Z, Masarova L, Sasaki K, Verstovsek S, Ferrajoli A, Weirda WG, Wang SA, Konoplev S, Chen Z, Pierce SA, Ning J, Qiao W, Ravandi F, Andreeff M, Welch JS, Kantarjian HM, Konopleva MY. 10-day decitabine with venetoclax for newly diagnosed intensive chemotherapy ineligible, and relapsed or refractory acute myeloid leukaemia: a single-centre, phase 2 trial. Lancet Haematol. 2020 Oct;7(10):e724-e736. doi: 10.1016/S2352-3026(20)30210-6. Epub 2020 Sep 5. PMID 32896301
- [Background] DiNardo CD, Lachowiez CA, Takahashi K, Loghavi S, Xiao L, Kadia T, Daver N, Adeoti M, Short NJ, Sasaki K, Wang S, Borthakur G, Issa G, Maiti A, Alvarado Y, Pemmaraju N, Montalban Bravo G, Masarova L, Yilmaz M, Jain N, Andreeff M, Jabbour E, Garcia-Manero G, Kornblau S, Ravandi F, Konopleva MY, Kantarjian HM. Venetoclax Combined With FLAG-IDA Induction and Consolidation in Newly Diagnosed and Relapsed or Refractory Acute Myeloid Leukemia. J Clin Oncol. 2021 Sep 1;39(25):2768-2778. doi: 10.1200/JCO.20.03736. Epub 2021 May 27. PMID 34043428